CLINICAL TRIAL: NCT05909618
Title: An Open Label Phase 2 Study of Intravenously Administered Crizanlizumab Alone or in Combination With Nivolumab for Glioblastoma and Melanoma With Brain Metastases
Brief Title: Crizanlizumab Alone or in Combination With Nivolumab for Glioblastoma and Melanoma With Brain Metastases
Acronym: 14
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Prof. Ronit Satchi-Fainaro, Director, Cancer Biology Research Center, Tel Aviv University, Tel Aviv, Israel. (Unknown)
Responsible Party: Principal Investigator, Dr. Ronnie Shapira, M.D, Head onco-gynecological service, Principal Investigator, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sheba-9411-22-RS-crizanlizumab
Record Dates: First submitted 2023-05-01; First posted 2023-06-18 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Advanced Glioblastoma; Metastatic Melanoma in the Central Nervous System; MGMT-Unmethylated Glioblastoma
MeSH Terms: interventions — crizanlizumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 metastatic melanoma with brain metastases who failed immunotherapy (Experimental): The first 3 subjects enrolled to Cohort 1 and Cohort 2 will receive crizanlizumab 5 mg/kg at Cycle 1 Day 1 (C1D1) and C1D15 followed by crizanlizumab 5 mg/kg every 4 weeks until disease progression The subsequent 8 patients will receive crizanlizumab 5 mg/kg at C1D1 and C1D15 followed by 5 mg/kg every 4 weeks plus nivolumab 3mg/kg every 2 weeks until disease progression
- Cohort 2 - Patients with recurrent or progressing GB following radiation and temozolamide. (Experimental): The first 3 subjects enrolled to Cohort 1 and Cohort 2 will receive crizanlizumab 5 mg/kg at Cycle 1 Day 1 (C1D1) and C1D15 followed by crizanlizumab 5 mg/kg every 4 weeks until disease progression The subsequent 8 patients will receive crizanlizumab 5 mg/kg at C1D1 and C1D15 followed by 5 mg/kg every 4 weeks plus nivolumab 3mg/kg every 2 weeks until disease progression
  Interventions: Drug: Crizanlizumab-Tmca 10 MG/1 ML Intravenous Solution [ADAKVEO]; Drug: Nivolumab 10 MG/1 ML Intravenous Solution [OPDIVO]
- Cohort 3: Patients with newly diagnosed GB (Experimental): crizanlizumab starting from 4 weeks after completing radiation therapy. The first 2 subjects will receive crizanlizumab 2.5 mg/kg at C1D1 and C1D15 followed by crizanlizumab 5 mg/kg every 4 weeks. The subsequent 6 subjects will receive crizanlizumab 5 mg/kg at C1D1 and C1D15 followed by crizanlizumab every 4 weeks. Treatment will continue for up to 12 months or until disease progression or unacceptable toxicity.
  Interventions: Drug: Crizanlizumab-Tmca 10 MG/1 ML Intravenous Solution [ADAKVEO]

INTERVENTIONS:
Drug: Crizanlizumab-Tmca 10 MG/1 ML Intravenous Solution [ADAKVEO] — 5 mg/kg solution for injection
  Other Names: crizanlizumab
  Arms: Cohort 2 - Patients with recurrent or progressing GB following radiation and temozolamide.; Cohort 3: Patients with newly diagnosed GB
Drug: Nivolumab 10 MG/1 ML Intravenous Solution [OPDIVO] — 3 mg/mL solution for injection
  Other Names: nivolumab
  Arms: Cohort 2 - Patients with recurrent or progressing GB following radiation and temozolamide.

SUMMARY:
A single-center, open-label, non-randomized phase I/II study to evaluate the efficacy, safety and tolerance of crizanlizumab monotherapy and in combination with nivolumab in patients with advanced glioblastoma (GB) who exhausted standard of care (SOC) therapy, patients with metastatic brain melanoma (MBM) and patients with newly diagnosed unmethylated GB.

Subjects will be screened for up to 28 days prior to treatment initiation. Eligible subjects will be allocated to one of 3 cohorts:

Cohort 1: Patients with metastatic melanoma with primarily diagnosed or newly progressing brain metastases who failed immunotherapy.

Cohort 2: Patients with recurrent or progressing GB following primary radiation therapy and temozolomide. Patients may have failed up to 2 prior systemic treatment lines (including temozolomide as adjuvant therapy) and are candidates for further treatment.

Cohort 3: Patients with newly diagnosed GB who were evaluated for methylguanine-DNA methyltransferase(MGMT) methylation status and have un-methylated MGMT promotor-therefore, they are not candidates for maintenance temozolomide therapy.

DETAILED DESCRIPTION:
A single-center, open-label, non-randomized phase I/II study to evaluate the efficacy, safety and tolerance of crizanlizumab monotherapy and in combination with nivolumab in patients with advanced glioblastoma (GB) who exhausted standard of care (SOC) therapy, patients with metastatic brain melanoma (MBM) and patients with newly diagnosed unmethylated GB.

Subjects will be screened for up to 28 days prior to treatment initiation. Eligible subjects will be allocated to one of 3 cohorts:

Cohort 1: Patients with metastatic melanoma with primarily diagnosed or newly progressing brain metastases who failed immunotherapy.

Cohort 2: Patients with recurrent or progressing GB following primary radiation therapy and temozolomide. Patients may have failed up to 2 prior systemic treatment lines (including temozolomide as adjuvant therapy) and are candidates for further treatment.

Cohort 3: Patients with newly diagnosed GB who were evaluated for MGMT methylation status and have un-methylated MGMT promotor-therefore, they are not candidates for maintenance temozolomide therapy.

The first 3 subjects enrolled to Cohort 1 and Cohort 2 will receive crizanlizumab 5 mg/kg at Cycle 1 Day 1 (C1D1) and Cycle 1 Day 15 (C1D15) followed by crizanlizumab 5 mg/kg every 4 weeks until disease progression evaluated by RECIST 1.1 and RANO criteria or intolerable toxicity. The subsequent 8 patients will receive crizanlizumab 5 miligram/kilogram (mg/kg) at C1D1 and C1D15 followed by 5 mg/kg every 4 weeks plus nivolumab 3mg/kg every 2 weeks until disease progression. The subjects will continue the treatment until disease progression or until completion of 27 cycles (2 years). Subjects who complete 2 years of therapy will maintain follow-up.

Subjects in Cohort 3 will receive crizanlizumab starting from 4 weeks after completing radiation therapy. The first 2 subjects will receive crizanlizumab 2.5 mg/kg at C1D1 and C1D15 followed by crizanlizumab 5 mg/kg every 4 weeks. The subsequent 6 subjects will receive crizanlizumab 5 mg/kg at C1D1 and C1D15 followed by crizanlizumab every 4 weeks. Treatment will continue for up to 12 months or until disease progression or unacceptable toxicity.

Safety and tolerability will be assessed by CTCAE v 6.0 every week for the first 4 weeks followed by assessments every 2 weeks until Week 12, and then every 4 weeks.

Tumor response will be evaluated by brain Magnetic resonance imaging (MRI) every 8 weeks using RANO criteria. Patients with metastatic melanoma will also be evaluated with chest-abdomen and pelvis Computed tomography (CT) every 8 weeks for the evaluation of visceral disease using RECIST 1.1.

Patients with MBM (Cohort 1) whose primary tumor/non-brain tumor progresses on RECIST 1.1 but whose brain tumor/metastases show benefit (stable disease or better), may continue in the study at the investigator's discretion.

Quality of life will be assessed by the Quality of Life Questionnaire (EORTC QLQ-30) and Brain Neoplasm(QLQ BN-20) and by cognitive function tests.

Archived tissue samples (and optional fresh biopsy), CSF and blood samples will be drawn to assess pharmacokinetics and pharmacodynamics of the combined therapy and for collateral research aiming to define biomarkers for response.

ELIGIBILITY:
Cohort 1 (MBM) Inclusion Criteria

1. Age ≥ 18 years.
2. Estimated life expectancy at least 3 months
3. Have metastatic melanoma with primarily diagnosed or newly progressing brain metastases.
4. Was treated with 1 prior systemic line of immunotherapy - either PD-1 inhibitor monotherapy or combined CTLA4 and PD-1 antibodies or another investigational combination of immunotherapy. Patients with BRAF-mutant melanoma who have also received BRAF mutation targeted therapy are also eligible.
5. Have failed prior immunotherapy line, either due to primary resistance or acquired resistance.
6. Have measurable disease defined by RECIST criteria and have at least one, non-previously irradiated brain metastasis of at least 1-cm short diameter. Otherwise, previously irradiated lesions should present with enlargement following radiation therapy.
7. Is clinically stable with no neurological deficits. Patients may receive steroid supportive therapy up to 10 mg of prednisone or the equivalent.
8. Have Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
9. Adequate organ function defined by blood tests for blood count and chemistry.
10. Women of childbearing potential practicing an acceptable method of birth control.
11. Understand study procedures and willingness to comply for the entire duration of the study and to give written informed consent.

    Exclusion Criteria
12. Systemic steroid therapy for symptomatic brain disease. Note: a dose equivalent to 10 mg prednisone will be allowed
13. Have leptomeningeal spread.
14. Previous life-threatening toxicity to anti-PD-1 antibody monotherapy.
15. Auto-immune disease in the last 2 years requiring systemic immune-suppressive therapy.
16. Previous exposure to Crizanlizumab or any other P-selectin inhibitor.
17. Previous or current brain hemorrhage.
18. The patient had, or is expected to undergo, allogeneic hematopoietic stem cell transplantation (HSCT).
19. The patient had a contraindication for undergoing brain MRI.
20. Any other severe concurrent disease which, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
21. Pregnant or lactating
22. Treatment with other investigational drugs within <21 days of start of day 1 of the study treatment.
23. Any contraindication for treatment with nivolumab according to the product's labels.

Cohort 2 (Recurrent or Progressive GB) Inclusion Criteria

1. Age ≥ 18 years.
2. Estimated life expectancy at least 3 months
3. Have with recurrent or persistent GB
4. Received first line therapy with brain irradiation and maintenance temozolamide.
5. Measurable disease per RANO criteria on brain MRI.
6. Have Eastern Cooperative Oncology Group (ECOG) performance status <2.
7. Adequate organ function defined by blood tests for blood count and chemistry.
8. Women of childbearing potential practicing an acceptable method of birth control.
9. Understand study procedures and willingness to comply for the entire duration of the study and to give written informed consent.

Exclusion Criteria

1. Systemic steroid therapy for symptomatic brain disease. Note: a dose equivalent to 20 mg prednisone will be allowed
2. Have leptomeningeal spread.
3. Previous life-threatening toxicity to anti-PD-1 antibody monotherapy.
4. Auto-immune disease in the last 2 years requiring systemic immune-suppressive therapy.
5. Previous exposure to Crizanlizumab or any other P-selectin inhibitor.
6. Previous or current brain hemorrhage.
7. The patient had, or is expected to undergo, allogeneic HSCT.
8. The patient had a contraindication for undergoing brain MRI.
9. Any other severe concurrent disease which, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
10. Pregnant or lactating
11. Treatment with other investigational drugs within <21 days of start of day 1 of the study treatment.
12. Any contraindication for treatment with nivolumab according to the product's labels.

Cohort 3 (Newly Diagnosed Unmethylated GB) Inclusion Criteria

1. Age ≥ 18 years.
2. Estimated life expectancy at least 3 months.
3. Histologically confirmed newly diagnosed GB.
4. Tumor test result shows MGMT unmethylated type.
5. Received definitive brain irradiation.
6. Patients may be treated with novo TTF (optune) per local standard.
7. Have Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
8. Adequate organ function defined by blood tests for blood count and chemistry.
9. Women of childbearing potential practicing an acceptable method of birth control.
10. Understand study procedures and willingness to comply for the entire duration of the study and to give written informed consent.

Exclusion Criteria

1. Systemic steroid therapy for symptomatic brain disease. Note: a dose equivalent to 20 mg prednisone will be allowed
2. Have leptomeningeal spread.
3. Previous life-threatening toxicity to anti-PD-1 antibody monotherapy.
4. Auto-immune disease in the last 2 years requiring systemic immune-suppressive therapy.
5. Previous exposure to Crizanlizumab or any other P-selectin inhibitor.
6. Previous or current brain hemorrhage.
7. The patient had, or is expected to undergo, allogeneic HSCT.
8. The patient had a contraindication for undergoing brain MRI.
9. Any other severe concurrent disease which, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
10. Be pregnant or lactating
11. Treatment with other investigational drugs within <21 days of start of day 1 of the study treatment.

Any contraindication for treatment with nivolumab according to the product's labels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2028-07-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse, serious adverse events, immune-related AEs following treatment with crizanlizumab alone or in combination with nivolumab | 48 months
  Safety and tolerability assessed by CTCAE v 6.0
The proportion of treatment discontinuation events related to the treatment combination | 48 months
  Safety and tolerability assessed by CTCAE v 6.0

SECONDARY OUTCOMES:
Response Rate (RR) to crizanlizumab monotherapy and in combination with nivolumab | 48 months
  evaluated by RECIST 1.1 and by RANO and RANO-BM criteria.
Progression-free survival (PFS) of patients with GB or MBM following treatment crizanlizumab monotherapy and in combination with nivolumab | evaluated every 8 weeks for 48 months
  by brain MRI and CT of chest/abdomen and pelvis using RECIST 1.1 and RANO/RANO-BM criteria
Overall survival (OS) in patients with GB or MBM following treatment crizanlizumab monotherapy and in combination with nivolumab. | 48 months
  Overall survival (OS) of the study population
Impact of the treatment protocol on health-related quality of life | evaluated every 6 weeks for 48 months
  using EORTC questionnaires ,All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Incidence of treatment-related adverse, serious adverse events, immune-related AEs of crizanlizumab maintenance therapy following whole-brain irradiation in patients with unmethylated GB | 48 months
  evaluated by adverse events monitoring using CTCAE Version 6.0 and by documenting study treatment discontinuation and delays.
Disease control rate (DCR) | 48 months
  valuated by rate of progression in patients with un-methylated GB treated with crizanlizumab maintenance therapy following whole-brain irradiation.

OTHER OUTCOMES:
The response to crizanlizumab monotherapy and in combination with nivolumab | 48 months
  by iRANO criteria
Plasma levels of Crizanlizumab measurements | during the first treatment cycle at the following time points: Baseline (Day 1),Day 2 and Day 15.
  Plasma levels of Crizanlizumab will be measured. The following parameters will be calculated: maximum (peak) plasma drug concentration (Cmax), area under the plasma concentration-time curve from time zero to time t (AUC0-t), area under the plasma concentration-time curve from time zero to infinity (AUC0-∞), mean residence time (MRT), elimination half-life (t½), elimination rate constant (Kel), apparent total body clearance of the drug from plasma (Cl), apparent volume of distribution (Vd).
  evaluated by blood for pharmacokinetics analyses that will be collected at the following time points:
  * Baseline (Day 1) prior to dosing and at 15 min, 30 min, 1 hour, 2 hours, 4 hours, and 8 ±1 hour post-dosing.
  * Day 2, at 20-24 hours post dosing.
  * Day 15±1 prior to dosing and at 15 min, 30 min, 1 hour, 2 hours, 4 hours, and 8 ±1 hour post-dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Shapira Frommer, Dr, Principal Investigator — Ronnie Shapira, MD Study Principal Investigator Ronnie.Shapira@sheba.health.gov.il
Locations (1):
- Sheba medical center, Ramat Gan, Israel, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Nature Communications manuscript — https://www.nature.com/articles/s41467-021-22186-0